CLINICAL TRIAL: NCT00040846
Title: Campath® [Alemtuzumab] Dose Escalation, Low-Dose TBI and Fludarabine Followed by HLA Class I Mismatched Donor Stem Cell Transplantation for Patients With Hematologic Malignancies - A Multi-Center Trial
Brief Title: Alemtuzumab, Fludarabine Phosphate, and Low-Dose Total Body Irradiation Before Donor Stem Cell Transplantation in Treating Patients With Hematological Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Brenda Sandmaier, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1591.00; NCI-2011-00471 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1591.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH); P01CA018029 (NIH)
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Results first posted 2017-03-16 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Childhood Burkitt Lymphoma; Childhood Chronic Myelogenous Leukemia; Childhood Diffuse Large Cell Lymphoma; Childhood Immunoblastic Large Cell Lymphoma; Childhood Nasal Type Extranodal NK/T-cell Lymphoma; Chronic Phase Chronic Myelogenous Leukemia; Contiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Contiguous Stage II Grade 1 Follicular Lymphoma; Contiguous Stage II Grade 2 Follicular Lymphoma; Contiguous Stage II Marginal Zone Lymphoma; Contiguous Stage II Small Lymphocytic Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Noncontiguous Stage II Grade 1 Follicular Lymphoma; Noncontiguous Stage II Grade 2 Follicular Lymphoma; Noncontiguous Stage II Marginal Zone Lymphoma; Noncontiguous Stage II Small Lymphocytic Lymphoma; Peripheral T-cell Lymphoma; Previously Treated Myelodysplastic Syndromes; Progressive Hairy Cell Leukemia, Initial Treatment; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Childhood Anaplastic Large Cell Lymphoma; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Recurrent/Refractory Childhood Hodgkin Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Refractory Multiple Myeloma; Relapsing Chronic Myelogenous Leukemia; Splenic Marginal Zone Lymphoma; Stage I Adult Diffuse Small Cleaved Cell Lymphoma; Stage I Childhood Anaplastic Large Cell Lymphoma; Stage I Childhood Large Cell Lymphoma; Stage I Cutaneous T-cell Non-Hodgkin Lymphoma; Stage I Grade 1 Follicular Lymphoma; Stage I Grade 2 Follicular Lymphoma; Stage I Mantle Cell Lymphoma; Stage I Marginal Zone Lymphoma; Stage I Mycosis Fungoides/Sezary Syndrome; Stage I Small Lymphocytic Lymphoma; Stage II Childhood Anaplastic Large Cell Lymphoma; Stage II Childhood Large Cell Lymphoma; Stage II Cutaneous T-cell Non-Hodgkin Lymphoma; Stage II Mycosis Fungoides/Sezary Syndrome; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Childhood Anaplastic Large Cell Lymphoma; Stage III Childhood Large Cell Lymphoma; Stage III Cutaneous T-cell Non-Hodgkin Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Mycosis Fungoides/Sezary Syndrome; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Childhood Anaplastic Large Cell Lymphoma; Stage IV Childhood Large Cell Lymphoma; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Mycosis Fungoides/Sezary Syndrome; Stage IV Small Lymphocytic Lymphoma; T-cell Large Granular Lymphocyte Leukemia; Waldenström Macroglobulinemia
MeSH Terms: conditions — Congenital Abnormalities; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Leukemia, Myeloid, Chronic-Phase; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence; Leukemia, Hairy Cell; Multiple Myeloma; Leukemia, Large Granular Lymphocytic; Waldenstrom Macroglobulinemia | interventions — Alemtuzumab; fludarabine phosphate; Whole-Body Irradiation; Peripheral Blood Stem Cell Transplantation; Mycophenolic Acid; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (dose-escalation of alemtuzumab, HSCT) (Experimental): CONDITIONING REGIMEN: Patients receive alemtuzumab IV over 2 hours on days -8 to -5 and fludarabine phosphate IV on days -4 to -2. Patients also undergo low-dose TBI on day 0.
  HSCT: Patients undergo allogeneic peripheral blood stem cell transplantation on day 0.
  IMMUNOSUPPRESSION: Patients receive CSP IV or PO BID on days -3 to 180 with taper to day 365 and MMF PO TID on days 0-100, with taper to day 156.
  Interventions: Biological: alemtuzumab; Drug: fludarabine phosphate; Radiation: total-body irradiation; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Drug: mycophenolate mofetil; Drug: cyclosporine

INTERVENTIONS:
Biological: alemtuzumab — Given IV
  Other Names: anti-CD52 monoclonal antibody; Campath-1H; MoAb CD52; Monoclonal Antibody Campath-1H; Monoclonal Antibody CD52
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Radiation: total-body irradiation — Undergo TBI
  Other Names: TBI
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo allogeneic HSCT
Procedure: peripheral blood stem cell transplantation — Undergo allogeneic peripheral blood stem cell transplantation
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Drug: mycophenolate mofetil — Given PO
  Other Names: Cellcept; MMF
Drug: cyclosporine — Given IV or PO
  Other Names: ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune

SUMMARY:
This phase II trial studies the side effects and the best dose of alemtuzumab when given together with fludarabine phosphate and low-dose total body irradiation (TBI) and how well it works before donor stem cell transplant in treating patients with hematological malignancies. Giving chemotherapy and low-dose TBI before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. Also, monoclonal antibodies, such as alemtuzumab, can find cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine (CSP) and mycophenolate mofetil (MMF) after transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether stable allogeneic engraftment from related and unrelated human leukocyte antigen (HLA)-mismatched stem cell donors can be safely established using a non-myeloablative conditioning regimen plus escalating doses of the anti-CD52 monoclonal antibody (mAb) Campath (alemtuzumab) in patients with hematologic malignancies.

SECONDARY OBJECTIVES:

I. Evaluate the risk of occurrence of acute and chronic graft-vs-host disease (GVHD).

II. Evaluate the risk/incidence of infections.

III. Determine whether engraftment can be maintained with a single dose fludarabine, donor lymphocyte infusion (DLI) and continued MMF/CSP.

IV. Evaluate the risk for disease progression and relapse.

OUTLINE: This is a dose-escalation study of alemtuzumab.

CONDITIONING REGIMEN: Patients receive alemtuzumab intravenously (IV) over 2 hours on days -8 to -5 and fludarabine phosphate IV on days -4 to -2. Patients also undergo low-dose TBI on day 0.

HEMATOPOIETIC STEM CELL TRANSPLANTATION (HSCT): Patients undergo allogeneic peripheral blood stem cell transplantation on day 0.

IMMUNOSUPPRESSION: Patients receive CSP IV or orally (PO) twice daily (BID) on days -3 to 180 with taper to day 365 and MMF PO thrice daily (TID) on days 0-100 with taper to day 156.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be not eligible for conventional transplants and must have disease expected to be stable for at least 100 days without chemotherapy; patients with hematologic malignancies treatable with hematopoietic stem cell transplant (HSCT) or with a B cell malignancy except those treatable with autologous transplant will be included
* Aggressive non-Hodgkin lymphomas (NHLs) and Other Histologies Such as Diffuse large B cell NHL

  * Patients with primary refractory or relapsed disease not eligible for an autologous transplant
  * Patients are eligible following an autologous transplant in remission or in relapse
  * Planned tandem transplant is allowed for patients at high risk of relapse
* Low grade NHL with < 6 months duration of complete remission (CR) between courses of conventional therapy
* Mantle Cell NHL may be treated in first CR
* Chronic lymphocytic leukemia (CLL) - Must have failed 2 lines of conventional therapy and be refractory to fludarabine
* Hodgkin disease (HD) - Must have received and failed frontline therapy; patients must have had a prior autologous transplant or were not eligible for autologous transplant; planned tandem transplants are allowed for patients at high risk of relapse
* Multiple myeloma (MM) - Must have received prior chemotherapy and a prior autologous transplant, unless autologous transplant was not possible; planned tandem transplants are allowed for patients at high risk of relapse
* Acute myeloid leukemia (AML) - Must have < 5% marrow blasts at the time of transplant
* Acute lymphocytic leukemia (ALL) - Must have < 5% blasts at the time of transplant
* Chronic myeloid leukemia (CML) - Patients will be accepted beyond chronic phase 1 (CP1) if they have received previous myelosuppressive chemotherapy or HSCT, and have < 5% marrow blasts at time of transplant
* Myelodysplastic (MDS)/Myeloproliferative disorders - Must have failed previous myelosuppressive chemotherapy or HSCT, and have < 5% marrow blasts at time of transplant
* Waldenstrom's Macroglobulinemia - Must have failed 2 courses of therapy
* Patients < 12 years old must be approved by the Fred Hutchinson Cancer Research Center (FHCRC) principal investigator (PI)
* Patients who refuse to be treated on a conventional transplant protocol; for this inclusion, criteria transplants must be approved by both the participating institution´s patient review committee such as the Patient Care Conference (PCC) at the FHCRC and the FHCRC principal investigator
* Patients with related or unrelated donors for whom

  * The best available match is a HLA class II DRB1 and DQB1 matched donor incompatible for any single serologically detectable class I HLA-A, -B, -C mismatch; one additional allele level class I mismatch is allowed OR any combination of 2 allele level mismatches (if typed at the molecular level)
  * There is a likelihood of rapid disease progression while HLA typing and results of a preliminary search and the donor pool suggests that a 10/10 HLA-A, B, C, DRB1 and DQB1 matched unrelated donor will not be found
  * There is no HLA-A, -B or -C one locus allelic mismatched related donor available
  * There is no indication for an autologous transplantation as a treatment option
* DONOR: Related or unrelated donors who are matched for HLA-DRB1 and DQB1 alleles (must be defined by high resolution typing), and who are mismatched for:

  * Any single serologically detectable HLA-A or B or C antigen +/- 1 allele or
  * Any combination of two HLA-A, -B, or -C alleles (if prospectively typed at molecular level)

Exclusion Criteria:

* Patients who are homozygous at the mismatched major histocompatibility complex (MHC) class I locus
* A positive cross-match exists between the donor and recipient
* Patients with rapidly progressive intermediate or high grade NHL
* Presence of circulating leukemic blasts (in the peripheral blood) detected by standard pathology for patients with AML, ALL or CML
* Life expectancy severely limited by diseases other than malignancy
* Central nervous system (CNS) involvement with disease refractory to intrathecal chemotherapy
* Fertile men or women unwilling to use contraceptives during and for up to 12 months post treatment
* Female patients who are pregnant or breast-feeding
* Human immunodeficiency virus (HIV) positive patients
* Patients with active non-hematologic malignancies (except non-melanoma skin cancers)
* Patients with a history of non-hematologic malignancies (except non-melanoma skin cancers) currently in a complete remission, who are less than 5 years from the time of complete remission, and have a > 20% risk of disease recurrence
* Fungal infections with radiological progression after receipt of amphotericin B or active triazole for greater than 1 month
* Patients with active bacterial or fungal infections unresponsive to medical therapy
* Patients with the following organ dysfunction symptomatic coronary artery disease or ejection fraction < 35% or other cardiac failure requiring therapy; ejection fraction is required if the patient is > 50 years of age, or history of cardiac disease or anthracycline exposure

  * Diffusion capacity of carbon monoxide (DLCO) < 35%; total lung capacity (TLC) < 35%; or forced expiratory volume in one second (FEV1) < 35% and/or receiving supplementary continuous oxygen
  * Patients with clinical or laboratory evidence of liver disease would be evaluated for the cause of liver disease, its clinical severity in terms of liver function, bridging fibrosis, and the degree of portal hypertension; patients will be excluded if they are found to have fulminant liver failure; cirrhosis of the liver with evidence of portal hypertension; alcoholic hepatitis; esophageal varices; a history of bleeding esophageal varices; hepatic encephalopathy; uncorrectable hepatic synthetic dysfunction evinced by prolongation of the prothrombin time; ascites related to portal hypertension; bacterial or fungal liver abscess; biliary obstruction; chronic viral hepatitis with total serum bilirubin >3 mg/dL; or symptomatic biliary disease
  * Patients with poorly controlled hypertension on multiple antihypertensives
  * Karnofsky score < 70 for adult patients
  * Lansky-Play Performance Score < 50 for pediatric patients
* DONOR: Bone marrow (BM) donors
* DONOR: Donors who are HIV-positive and/or, medical conditions that would result in increased risk for granulocyte colony-stimulating factor (G-CSF) mobilization and harvest of peripheral blood stem cell (PBSC)
* DONOR: Donors < 12 years of age

Max Age: 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2001-11 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Sandmaier, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (7):
- United States (6):
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - VA Puget Sound Health Care System, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Froedtert Memorial Lutheran Hospital, Medical College of Wisconsin, Milwaukee, Wisconsin
- University of Torino, Torino, Italy

REFERENCES:
- [Result] Nakamae H, Storer BE, Storb R, Storek J, Chauncey TR, Pulsipher MA, Petersen FB, Wade JC, Maris MB, Bruno B, Panse J, Petersdorf E, Woolfrey A, Maloney DG, Sandmaier BM. Low-dose total body irradiation and fludarabine conditioning for HLA class I-mismatched donor stem cell transplantation and immunologic recovery in patients with hematologic malignancies: a multicenter trial. Biol Blood Marrow Transplant. 2010 Mar;16(3):384-94. doi: 10.1016/j.bbmt.2009.11.004. Epub 2009 Nov 10. PMID 19900571

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1 (No Campath): CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV on days -4 to -2. Patients also undergo low-dose TBI on day 0.
  HSCT: Patients undergo allogeneic peripheral blood stem cell transplantation on day 0.
  IMMUNOSUPPRESSION: Patients receive CSP IV or PO BID on days -3 to 180 with taper to day 365 and MMF PO TID on days 0-100, with taper to day 156.
  fludarabine phosphate: Given IV
  total-body irradiation: Undergo TBI
  allogeneic hematopoietic stem cell transplantation: Undergo allogeneic HSCT
  peripheral blood stem cell transplantation: Undergo allogeneic peripheral blood stem cell transplantation
  mycophenolate mofetil: Given PO
  cyclosporine: Given IV or PO
- Dose Level 2 (0.025 mg/kg/Day Campath); Dose Level 3 (0.050 mg/kg/Day Campath); Dose Level 4 (0.10 mg/kg/Day Campath); Dose Level 5 (0.20 mg/kg/Day Campath); Dose Level 6 (0.40 mg/kg/Day Campath): CONDITIONING REGIMEN: Patients receive Alemtuzumab (Campath) on days -8 to -5 as well as fludarabine phosphate IV on days -4 to -2. Patients also undergo low-dose TBI on day 0.
  HSCT: Patients undergo allogeneic peripheral blood stem cell transplantation on day 0.
  IMMUNOSUPPRESSION: Patients receive CSP IV or PO BID on days -3 to 180 with taper to day 365 and MMF PO TID on days 0-100, with taper to day 156.
  fludarabine phosphate: Given IV
  total-body irradiation: Undergo TBI
  allogeneic hematopoietic stem cell transplantation: Undergo allogeneic HSCT
  peripheral blood stem cell transplantation: Undergo allogeneic peripheral blood stem cell transplantation
  mycophenolate mofetil: Given PO
  cyclosporine: Given IV or PO
  alemtuzumab: Given IV
Period: Overall Study
Arm/Group | Dose Level 1 (No Campath) | Dose Level 2 (0.025 mg/kg/Day Campath) | Dose Level 3 (0.050 mg/kg/Day Campath) | Dose Level 4 (0.10 mg/kg/Day Campath) | Dose Level 5 (0.20 mg/kg/Day Campath) | Dose Level 6 (0.40 mg/kg/Day Campath)
Started | 60 | 0 | 0 | 0 | 0 | 0
Completed | 60 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No subjects were enrolled onto groups beyond Dose level 1 because the dose escalation was not triggered over the course of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 (No Campath) | Dose Level 2 (0.025 mg/kg/Day Campath) | Dose Level 3 (0.050 mg/kg/Day Campath) | Dose Level 4 (0.10 mg/kg/Day Campath) | Dose Level 5 (0.20 mg/kg/Day Campath) | Dose Level 6 (0.40 mg/kg/Day Campath) | Total
Number analyzed (Participants) | 60 | 0 | 0 | 0 | 0 | 0 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 |  |  |  |  |  | 1
  Between 18 and 65 years | 52 |  |  |  |  |  | 52
  >=65 years | 7 |  |  |  |  |  | 7
Age, Continuous [Median (Full Range); unit: years] | 56.7 [13 to 72] |  |  |  |  |  | 56.7 [13 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 |  |  |  |  |  | 15
  Male | 45 |  |  |  |  |  | 45
Region of Enrollment [Number; unit: participants]
  United States | 60 |  |  |  |  |  | 60

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Risk of Transplant Related Mortality.
Description: Percentage patients with Day 100 transplant related mortality.
Time Frame: 100 days after transplant
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Dose Level 1 (No Campath) | Dose Level 2 (0.025 mg/kg/Day Campath) | Dose Level 3 (0.050 mg/kg/Day Campath) | Dose Level 4 (0.10 mg/kg/Day Campath) | Dose Level 5 (0.20 mg/kg/Day Campath) | Dose Level 6 (0.40 mg/kg/Day Campath)
Number analyzed (Participants) | 60 | 0 | 0 | 0 | 0 | 0
percentage of participants | 20 |  |  |  |  |

2. Primary Outcome: Evaluate the Risk of Occurrence of Acute and Chronic GVHD
Description: Percentage patients who developed acute/chronic GVHD.
  aGVHD Stages
  Skin:
  1. a maculopapular eruption involving < 25% BSA
  2. a maculopapular eruption involving 25 - 50% BSA
  3. generalized erythroderma
  4. generalized erythroderma with bullous formation and often with desquamation
  Liver:
  1. bilirubin 2.0 - 3.0 mg/100 mL
  2. bilirubin 3 - 5.9 mg/100 mL
  3. bilirubin 6 - 14.9 mg/100 mL
  4. bilirubin > 15 mg/100 mL
  Gut:
  Diarrhea is graded 1 - 4 in severity. Nausea and vomiting and/or anorexia caused by GVHD is assigned as 1 in severity. The severity of gut involvement is assigned to the most severe involvement noted. Patients with visible bloody diarrhea are at least stage 2 gut and grade 3 overall.
  aGVHD Grades Grade III: Stage 2 - 4 gastrointestinal involvement and/or +2 to +4 liver involvement, with or without a rash Grade IV: Pattern and severity of GVHD similar to grade 3 with extreme constitutional symptoms or death
Time Frame: 1 year after transplant
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Dose Level 1 (No Campath) | Dose Level 2 (0.025 mg/kg/Day Campath) | Dose Level 3 (0.050 mg/kg/Day Campath) | Dose Level 4 (0.10 mg/kg/Day Campath) | Dose Level 5 (0.20 mg/kg/Day Campath) | Dose Level 6 (0.40 mg/kg/Day Campath)
Number analyzed (Participants) | 60 | 0 | 0 | 0 | 0 | 0
percentage of participants
  Grade III-IV aGVHD | 23.3 |  |  |  |  |
  cGVHD | 41.7 |  |  |  |  |

3. Primary Outcome: Determine Whether Engraftment Can be Maintained With a Single Dose Fludarabine, DLI and Continued MMF/CSP, Defined as Rejection Rate < 20%.
Description: Mixed chimerism will be defined as the detection of donor T cells (CD3+) and granulocytes (CD 33+), as a proportion of the total T cell and granulocyte population, respectively, of greater than 5% and less than 95% in the peripheral blood. Full donor chimerism is defined as > 95% donor CD3+ T cells.
Time Frame: 100 days after transplant
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Dose Level 1 (No Campath) | Dose Level 2 (0.025 mg/kg/Day Campath) | Dose Level 3 (0.050 mg/kg/Day Campath) | Dose Level 4 (0.10 mg/kg/Day Campath) | Dose Level 5 (0.20 mg/kg/Day Campath) | Dose Level 6 (0.40 mg/kg/Day Campath)
Number analyzed (Participants) | 60 | 0 | 0 | 0 | 0 | 0
percentage of participants
  CD3 - Graft rejection | 3.3 |  |  |  |  |
  CD3 - Mixed chimerism | 18.3 |  |  |  |  |
  CD3 - Full donor chimerism | 70 |  |  |  |  |
  CD3 - Unknown | 8.33 |  |  |  |  |
  CD33 - Graft Rejection | 1.7 |  |  |  |  |
  CD33 - Mixed chimerism | 3.3 |  |  |  |  |
  CD33 - Full donor chimerism | 80 |  |  |  |  |
  CD33 - Unknown | 15 |  |  |  |  |

4. Secondary Outcome: Evaluate the Risk/Incidence of Infections
Description: Percentage patients who experienced infections within 100 days post-transplant.
Time Frame: 100 days after transplant
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Dose Level 1 (No Campath) | Dose Level 2 (0.025 mg/kg/Day Campath) | Dose Level 3 (0.050 mg/kg/Day Campath) | Dose Level 4 (0.10 mg/kg/Day Campath) | Dose Level 5 (0.20 mg/kg/Day Campath) | Dose Level 6 (0.40 mg/kg/Day Campath)
Number analyzed (Participants) | 60 | 0 | 0 | 0 | 0 | 0
percentage of participants | 91.7 |  |  |  |  |

5. Secondary Outcome: Evaluate the Risk for Disease Progression and Relapse
Description: Percentage patients who relapsed/progressed within 1 year post-transplant.
Time Frame: 1 year after transplant
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Dose Level 1 (No Campath) | Dose Level 2 (0.025 mg/kg/Day Campath) | Dose Level 3 (0.050 mg/kg/Day Campath) | Dose Level 4 (0.10 mg/kg/Day Campath) | Dose Level 5 (0.20 mg/kg/Day Campath) | Dose Level 6 (0.40 mg/kg/Day Campath)
Number analyzed (Participants) | 60 | 0 | 0 | 0 | 0 | 0
percentage of participants | 21.7 |  |  |  |  |

ADVERSE EVENTS:
Time Frame: AEs: Conditioning through Day 100; SAEs: Conditioning through Day 200
Description: No subjects were enrolled onto groups beyond Dose level 1 because the dose escalation was not triggered over the course of the study.
Arm/Group | Dose Level 1 (No Campath) | Dose Level 2 (0.025 mg/kg/Day Campath) | Dose Level 3 (0.050 mg/kg/Day Campath) | Dose Level 4 (0.10 mg/kg/Day Campath) | Dose Level 5 (0.20 mg/kg/Day Campath) | Dose Level 6 (0.40 mg/kg/Day Campath)
Serious Adverse Events (participants affected / at risk) | 24/60 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 33/60 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (No Campath) (N=60) | Dose Level 2 (0.025 mg/kg/Day Campath) (N=0) | Dose Level 3 (0.050 mg/kg/Day Campath) (N=0) | Dose Level 4 (0.10 mg/kg/Day Campath) (N=0) | Dose Level 5 (0.20 mg/kg/Day Campath) (N=0) | Dose Level 6 (0.40 mg/kg/Day Campath) (N=0)
Cardiac troponin I increased (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GVHD (Immune system disorders) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (No Campath) (N=60) | Dose Level 2 (0.025 mg/kg/Day Campath) (N=0) | Dose Level 3 (0.050 mg/kg/Day Campath) (N=0) | Dose Level 4 (0.10 mg/kg/Day Campath) (N=0) | Dose Level 5 (0.20 mg/kg/Day Campath) (N=0) | Dose Level 6 (0.40 mg/kg/Day Campath) (N=0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other (Coagulopathy) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 13 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other (Blood) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Gram negative bacteremia, resulting in death
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infaction (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart Failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood and lymphatic System Disorder - Other (Hemoptysis) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other (BUN increased) (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes